CLINICAL TRIAL: NCT03519464
Title: A Phase 2, Open-Label Study to Assess the Immunogenicity of the 9-Valent Human Papillomavirus Recombinant Vaccine in Patients With Idiopathic CD4 T Cell Lymphocytopenia
Brief Title: Immunogenicity of the 9-Valent Human Papillomavirus Recombinant Vaccine in People With Idiopathic CD4 T Cell Lymphocytopenia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 180092; 18-I-0092
Record Dates: First submitted 2018-05-08; First posted 2018-05-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12-03

CONDITIONS: Idiopathic CD4 T Cell Lymphocytopenia
Keywords: Gardasil 9; Seroconversion; Humoral immune response; Cellular Immune Response; Mucosal Lesions
MeSH Terms: conditions — HIV Seropositivity | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ICL and Healthy Volunteers (Other): Biological/Vaccine
  Interventions: Biological: Gardasil 9

INTERVENTIONS:
Biological: Gardasil 9 — Gardasil 9 administered as a 0.5ml intramuscular injection in the deltoid region of the upper arm or in the anterolateral area of the thigh, 3-dose regimen of injections given at month 0, month 2, and month 6.

SUMMARY:
Background:

Diseases related to human papillomavirus (HPV) include warts, lesions, and cancers. ICL is idiopathic CD4 T cell lymphocytopenia. People with this rare disease get more HPV-related diseases than other people do. The diseases are more severe and harder to treat in people with ICL. Researchers want to see if the vaccine GARDASIL 9 can help people with ICL.

Objective:

To study the effects of the vaccine GARDASIL 9 in people with ICL.

Eligibility:

Adults ages 18-65 with ICL

Healthy volunteers the same age

Design:

Participants will be screened with a physical exam, medical history, and blood and pregnancy tests.

Participants will have a baseline visit with:

* Physical exam
* Medical history
* Oral rinse collection. Participants will gargle a small amount of a saline solution, then spit it into a cup.
* Apheresis. Blood will be removed through a needle in an arm. A machine will separate the blood and keep some parts for research. The rest will be returned to the participant through a needle in the other arm.
* Examination for HPV-related disease. Female participants will have a Pap test.

Researchers will collect swabs from some participants skin or genital lesions.

Participants will get 3 doses of the study vaccine over 6 months as a shot in the upper arm or thigh muscle. They will repeat the screening tests each vaccine visit.

Participants will record their temperature and side effects for several days after vaccinations.

Participants may have visits after vaccinations.

Participants will have 2 follow-up visits in the 18 months after the last vaccine. They will repeat most of the baseline tests.

...

DETAILED DESCRIPTION:
As observed in other immunocompromised individuals with selective or combined T cell deficits, the prevalence and morbidity of human papillomavirus (HPV)-related disease is increased in patients with idiopathic CD4 T cell lymphocytopenia (ICL). The high burden and aggressive clinical course of HPV-associated disease in patients with ICL requires the development of effective preventive measures in this specific population. The protection from a broader range of HPV types offered by the 9-valent vaccine is expected to be particularly beneficial in this population. This applies even to patients with a history of type-specific HPV-associated disease, as this population may remain at a higher risk of acquisition of infection with new oncogenic HPV types even with increasing age. However, the immunogenicity of vaccines and in particular HPV preventive vaccines has never been systematically studied in patients with ICL.

This will be a phase 2, open-label study to assess the immunogenicity of the U.S. Food and Drug Administration (FDA)-approved 9-valent HPV recombinant vaccine GARDASIL 9 in patients 18- through 70-years-old with ICL, irrespective of HPV serostatus, presence of HPV-associated diseases, or previous immunization with bivalent or quadrivalent HPV vaccine, as well as healthy controls matched to the ICL patient group for age and gender. The study will take place at a single site (National Institutes of Health Clinical Center, Bethesda, MD). Participants will be assessed at baseline for history and/or clinical evidence of HPV-associated disease. Those with a history of or current HPV skin or mucosal disease will undergo clinically indicated evaluation and be referred for clinical care as needed. We will administer the vaccine in a population of ICL patients ranging in age from 18 through 70 years old according to the standard 3-dose schedule approved by the FDA for individuals 9 through 45 years of age, with the second and third doses administered at least 2 months and at least 6 months, respectively, after the first dose. Follow-up visits will occur 1 and 18 months after completion of the vaccination schedule. Blood will be collected at each study visit for safety and immunogenicity testing.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged 18 to 70 years.
  2. Able to provide informed consent.
  3. Female study participants who engage in sexual activities that can result in pregnancy must agree to use one of the contraceptive methods listed below at every potentially reproductive sexual encounter, beginning at the baseline visit and continuing until 3 months after discontinuation of the study agent. Acceptable methods are as follows:
* Male or female condom with spermicide.
* Hormonal (e.g., consistent use of oral contraceptive pill daily or other hormonal method such as contraceptive implant or injection). Hormonal methods must be started 1 month prior to receiving the first dose of study agent.
* Diaphragm or cervical cap.
* Intrauterine device (IUD).

  4. Must meet criteria for 1 of the 2 study groups, as follows:
* Patients with ICL must have:

  * documented ICL, defined as CD4 cell count < 300 cells/microL in at least 2 different measurements 6 weeks apart, at any point in the past; and
  * CD4 cell count < 300 cells/microL (within 90 days prior to day 0, outside labs will be accepted).
  * If patient has documented ICL as defined in i. and is currently enrolled in NIH ICL natural history protocol (EPIC 09-I-0102) a CD4 cell count < 300 cells/ L (within 18 months of day 0) is sufficient for enrollment.
* Healthy volunteers must have:

  * CD4 cell count of greater than or equal to 450 cells/MicroL (within 90 days prior to day 0, outside labs will be accepted).

EXCLUSION CRITERIA:

1. Prior receipt of GARDASIL 9 (Receipt of 2-valent and 4-valent versions of vaccine is not exclusionary).
2. Pregnancy or breastfeeding.
3. History of hypersensitivity, including severe reactions to yeast or other component of the vaccine or to a previous vaccination with another GARDASIL vaccine.
4. HIV infection or any other recognized congenital or acquired immunodeficiency (i.e., SCID IL-2/JAK3/ADA, MAGT1, MHC1 deficiency, DOCK8, etc).
5. Current moderate or severe acute illness (i.e., febrile illness, seizure, myocardial infarction, cerebrovascular accident, pulmonary embolism) that in the opinion of the PI, would make the subject unsuitable for the study.
6. Serum creatinine > 1.5 times upper limit of normal, platelets < 100,0000/mm3, hemoglobin < 9 g/dL, or AST/ALT > 2 times upper limit of normal, immunoglobulin G level < 450 mg/liter.
7. Current use of systemic glucocorticosteroids or immunomodulants, other than corticosteroid nasal spray or inhaler and topical steroids, which are not exclusionary.
8. Any cancer diagnosis or autoimmune condition requiring systemic chemotherapy or immunomodulant affecting antibody responses (i.e., rituximab, ibrutinib etc.), intravenous or subcutaneous immunoglobulin supplementation, radiation therapy, or immunomodulatory treatment within the previous 6 months (presence of precancerous lesions is not exclusionary
9. Receipt of an investigational vaccine within 2 weeks of day 0.
10. Receipt of ACIP recommended immunizations within 1 week of day 0.
11. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with ICL who become seropositive to at least 1 homologous HPV vaccine genotype at 1 month after completion of the vaccination schedule. | 1 month (+ 1 month) after vaccination #3.
  Primary Endpoint: Proportion of patients with ICL who become seropositive to at least 1 homologous HPV vaccine genotype at 1 month after completion of the vaccination schedule.

SECONDARY OUTCOMES:
Humoral responses, expressed as geometric mean titer (GMT), will be compared between patients with ICL and healthy subjects, within the subgroup of subjects who seroconvert for any specific homologous HPV genotype. | 18 months after vaccination No 3.
  Secondary endpoint: Humoral responses, expressed as geometric mean titer (GMT), will be compared between patients with ICL and healthy subjects, within the subgroup of subjects who seroconvert for any specific homologous HPV genotype.
Number of adverse events (AEs) and serious adverse events (SAEs) following administration of 9-valent HPV recombinant vaccine. | 1 month (+ 1 month) after vaccination No3.
  Secondary endpoint: Number of adverse events (AEs) and serious adverse events (SAEs) following administration of 9-valent HPV recombinant vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lisco, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available at this time.

REFERENCES:
- [Background] Joura EA, Giuliano AR, Iversen OE, Bouchard C, Mao C, Mehlsen J, Moreira ED Jr, Ngan Y, Petersen LK, Lazcano-Ponce E, Pitisuttithum P, Restrepo JA, Stuart G, Woelber L, Yang YC, Cuzick J, Garland SM, Huh W, Kjaer SK, Bautista OM, Chan IS, Chen J, Gesser R, Moeller E, Ritter M, Vuocolo S, Luxembourg A; Broad Spectrum HPV Vaccine Study. A 9-valent HPV vaccine against infection and intraepithelial neoplasia in women. N Engl J Med. 2015 Feb 19;372(8):711-23. doi: 10.1056/NEJMoa1405044. PMID 25693011
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] Kumar D, Unger ER, Panicker G, Medvedev P, Wilson L, Humar A. Immunogenicity of quadrivalent human papillomavirus vaccine in organ transplant recipients. Am J Transplant. 2013 Sep;13(9):2411-7. doi: 10.1111/ajt.12329. Epub 2013 Jul 9. PMID 23837399
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0092.html